CLINICAL TRIAL: NCT01650805
Title: A Phase 3 Randomized,Open-Label Study of Ponatinib Versus Imatinib in Adult Patients With Newly Diagnosed Chronic Myeloid Leukemia in Chronic Phase
Brief Title: Ponatinib in Newly Diagnosed Chronic Myeloid Leukemia (CML) (EPIC)
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Study terminated based on evaluation of safety data.
Sponsor: Ariad Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AP24534-12-301
Expanded Access: NCT01592136 (Approved for marketing)
Record Dates: First submitted 2012-07-18; First posted 2012-07-26 (Estimated); Results first posted 2014-10-21 (Estimated); Last update posted 2014-11-17 (Estimated); Status verified 2014-10

CONDITIONS: Chronic Myeloid Leukemia
Keywords: Leukemia; Leukemia, Myeloid; Leukemia, Myelogenous, Chronic, BCR-ABL Positive; Neoplasms by Histologic Type; Neoplasms; Lymphoproliferative Disorders; Lymphatic Diseases; Immunoproliferative Disorders; Immune System Diseases; Myeloproliferative Disorders; Bone Marrow Diseases; Hematologic Diseases
MeSH Terms: conditions — Leukemia, Myelogenous, Chronic, BCR-ABL Positive; Leukemia; Leukemia, Myeloid; Neoplasms by Histologic Type; Neoplasms; Lymphoproliferative Disorders; Lymphatic Diseases; Immunoproliferative Disorders; Immune System Diseases; Myeloproliferative Disorders; Bone Marrow Diseases; Hematologic Diseases | interventions — ponatinib; Imatinib Mesylate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ponatinib (Experimental)
  Interventions: Drug: ponatinib
- imatinib (Active Comparator)
  Interventions: Drug: imatinib (Gleevec/ Glivec)

INTERVENTIONS:
Drug: ponatinib — 45 mg tablet, taken orally once daily
  Arms: ponatinib
Drug: imatinib (Gleevec/ Glivec) — 400 mg tablet, taken orally once daily
  Arms: imatinib

SUMMARY:
The purpose of this study is to compare the efficacy of ponatinib and imatinib in patients with newly diagnosed chronic myeloid leukemia (CML) in the chronic phase.

DETAILED DESCRIPTION:
This multicenter, international, phase 3 trial will test the hypothesis that ponatinib is an effective treatment for newly diagnosed CP-CML patients when compared with standard imatinib.

Patients will be randomized in a 1:1 fashion, stratified by Sokal risk score at diagnosis (low, intermediate, high), to receive once daily oral administration of either ponatinib or imatinib. Efficacy measures include molecular, cytogenetic, and hematologic response rates at various timepoints; time to, duration of, and durability of responses; and survival follow-up. Safety measures include clinical laboratory testing, adverse event monitoring, vital signs, physical exams, ECGs, and ECHOs. Other measures include two patient-reported health outcomes questionnaires (FACT-Leu and EQ-5D-5L), determination of mutation status, and, for ponatinib only, measurement of steady-state plasma concentration. Accrual is expected to take approximately 2 years, and patients will be followed for survival for up to 8 years after the last patient's first dose; therefore, patient participation may last up to 10 years.

ELIGIBILITY:
Inclusion Criteria:

1. CP CML within 6 months of diagnosis

   * CP-CML will be defined by (i) <15% blasts in bone marrow; (ii) <30% blasts plus promyelocytes in bone marrow; (iii) <20% basophils in peripheral blood; (iv) ≥100 × 10^9/L platelets (≥100,000/mm^3); (v) No evidence of extramedullary disease except hepatosplenomegaly; AND (vi) No prior diagnosis of AP-CML or BP-CML
2. Cytogenetic assessment must demonstrate the BCR-ABL fusion by presence of the t(9;22) Philadelphia chromosome

   * (a)Variant translocations are only allowed provided they are assessable for cytogenetic response utilizing conventional cytogenetic techniques; (b) Conventional chromosome banding must be performed; AND (c) A minimum of 20 metaphases must be assessable at entry
3. Eastern Cooperative Oncology Group (ECOG) Performance Status of 0, 1, or 2
4. Adequate hepatic function as defined by the following criteria:

   (a) Total serum bilirubin ≤1.5 x upper limit of normal (ULN), unless due to Gilbert's syndrome; (b) Alanine aminotransferase (ALT) ≤2.5 × ULN; AND (c) Aspartate aminotransferase (AST) ≤2.5 × ULN
5. Adequate renal function as defined as defined by serum creatinine <1.5 x ULN
6. Adequate pancreatic function as defined by serum lipase and amylase ≤1.5 × ULN

Exclusion Criteria:

1. Received prior imatinib therapy
2. Received prior dasatinib therapy
3. Received prior nilotinib therapy
4. Received, for CML, any other systemic anticancer therapy, experimental therapy, or radiation therapy with the exception of anagrelide or hydroxyurea
5. Major surgery within 28 days prior to initiating therapy
6. History of bleeding disorder unrelated to CML
7. History of acute pancreatitis within 1 year of study or history of chronic pancreatitis
8. History of alcohol abuse
9. Have uncontrolled hypertriglyceridemia (triglycerides >450 mg/dL)
10. Clinically significant, uncontrolled, or active cardiovascular disease, specifically including, but not restricted to:

    1. Myocardial infarction, within 6 months prior to randomization
    2. Unstable angina within 6 months prior to randomization
    3. Congestive heart failure within 6 months prior to randomization
    4. History of clinically significant (as determined by the treating physician) atrial arrhythmia or any ventricular arrhythmia
    5. Any history of ventricular arrhythmia
    6. Cerebrovascular accident or transient ischemic attack within 6 months prior to randomization
    7. Any history of peripheral arterial occlusive disease requiring revascularization
    8. Any history of venous thromboembolism including deep venous thrombosis or pulmonary embolism
11. Uncontrolled hypertension (diastolic blood pressure >90 mm Hg; systolic >140 mm Hg). Patients with hypertension should be under treatment on study entry to effect blood pressure control
12. Taking medications that are known to be associated with Torsades de Pointes
13. Ongoing or active infection. The requirement for intravenous (IV) antibiotics is considered active infection
14. Known history of human immunodeficiency virus (HIV). Testing is not required in the absence of history
15. Pregnant or breastfeeding
16. Malabsorption syndrome or other gastrointestinal illness that could affect oral absorption of study drugs
17. Diagnosed with or received anticancer therapy for another primary malignancy within 3 years prior to entry (except for non-melanoma skin cancer or cervical cancer in situ)
18. Any condition or illness that, in the opinion of the Investigator, would compromise patient safety or interfere with the evaluation of the drug

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 307 (Actual)
Dates: Start 2012-06; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

CONTACTS AND LOCATIONS:
Locations (170):
- United States (67):
  - US Oncology - Providence Health System, Site #167, Burbank, California
  - UCLA Department of Medicine, Site #027, Los Angeles, California
  - Bay Area Cancer Research Group, Site #156, Pleasant Hill, California
  - Bay Area Cancer Research Group, Site #157, Pleasant Hill, California
  - Rocky Mountain Cancer Centers, Site #191, Boulder, Colorado
  - Cancer Center of Central Connecticut, Site #147, Southington, Connecticut
  - Christiana Care Health Services, Site #155, Newark, Delaware
  - University Cancer Institute, Site #149, Boynton Beach, Florida
  - Florida Cancer Specialists, Site #180, Fort Meyers, Florida
  - Florida Cancer Specialists, Site #179, St. Petersburg, Florida
  - Emory University, Site #058, Atlanta, Georgia
  - John H. Stroger, Jr. Hospital of Cook County, Site #192, Chicago, Illinois
  - University of Chicago, Site #001, Chicago, Illinois
  - Loyola University Chicago, Site #054, Maywood, Illinois
  - Franciscan St. Francis Health, Site #138, Indianapolis, Indiana
  - University of Iowa Hospitals and Clinics, Site #050, Iowa City, Iowa
  - Siouxland Hematology-Oncology Associates, Site #198, Sioux City, Iowa
  - US Oncology - Cancer Center of Kansas, Site #168, Wichita, Kansas
  - Willis-Knighton Cancer Center, Site #196, Shreveport, Louisiana
  - University of Maryland, Greenebaum Cancer Center, Site #040, Baltimore, Maryland
  - Greater Baltimore Medical Center, Site #140, Baltimore, Maryland
  - St. Agnes Healthcare, Site #185, Baltimore, Maryland
  - Massachusetts General Hospital, Site #047, Boston, Massachusetts
  - Dana Farber Cancer Institute, Site #008, Boston, Massachusetts
  - University of Massachusetts Worcester, Site #152, Worcester, Massachusetts
  - University of Michigan Medical Center, Site #011, Ann Arbor, Michigan
  - Providence Cancer Institute, Site #197, Southfield, Michigan
  - Mayo Clinic, Site #044, Rochester, Minnesota
  - Oncology Research Park Nicollet Institute, Site #195, Saint Louis Park, Minnesota
  - Saint Luke's Hospital, Site #162, Kansas City, Missouri
  - Mercy Clinic - Cancer & Hematology, Site #151, Springfield, Missouri
  - Nebraska Hematology-Oncology, P.C., Site # 133, Lincoln, Nebraska
  - US Oncology - Comprehensive Cancer Center of Nevada, Site #169, Las Vegas, Nevada
  - John Theurer Cancer Center, Site #128, Hackensack, New Jersey
  - University of New Mexico Cancer Center, Site #166, Albuquerque, New Mexico
  - Maimonides Cancer Center, Site #177, Brooklyn, New York
  - Winthrop University Hospital, Site #153, Mineola, New York
  - Beth Israel Medical Center, Site #145, New York, New York
  - Mount Sinai School of Medicine, Site #189, New York, New York
  - Memorial Sloan-Kettering Cancer Center, Site #078, New York, New York
  - Weill Cornell Medical College, Site #006, New York, New York
  - New York Medical College, Site #146, Valhalla, New York
  - Southeastern Medical Oncology Center, Site #188, Goldsboro, North Carolina
  - Signal Point Clinical Research Center, Site #139, Middletown, Ohio
  - University of Oklahoma, Site #028, Oklahoma City, Oklahoma
  - Providence Cancer Center Oncology and Hematology Care Eastside, Site #194, Portland, Oregon
  - Kaiser Permanente Northwest, Site #200, Portland, Oregon
  - Oregon Health & Science University, Site #048, Portland, Oregon
  - Gettysburg Cancer Center, Site #160, Gettysburg, Pennsylvania
  - Western Pennsylvania Hospital, Site #159, Pittsburgh, Pennsylvania
  - Medical University of South Carolina, Site #148, Charleston, South Carolina
  - Carolina Hematology Oncology, Site #143, Sumter, South Carolina
  - Associates in Oncology & Hematology, Site #186, Chattanooga, Tennessee
  - Sarah Cannon Research Institute, Site #076, Nashville, Tennessee
  - US Oncology - Texas Oncology Austin, Site #172, Austin, Texas
  - US Oncology - Texas Oncology Dallas, Site #171, Dallas, Texas
  - University of Texas Southwestern Medical Center, Site #178, Dallas, Texas
  - Baylor College of Medicine, Site #063, Houston, Texas
  - US Oncology - Texas Oncology Midland, Site #173, Midland, Texas
  - US Oncology - Cancer Care Center of South Texas, Site #170, San Antonio, Texas
  - Huntsman Cancer Institute, Site #043, Salt Lake City, Utah
  - VCU Massey Cancer Center, Dalton Oncology Clinic, Site #069, Richmond, Virginia
  - Seattle Cancer Care Alliance, Site #100, Seattle, Washington
  - US Oncology - Northwest Cancer Specialists, Site #174, Vancouver, Washington
  - West Virginia University, Site #154, Morgantown, West Virginia
  - Green Bay Oncology, Ltd. / St. Mary's Hospital Medical Center, Site #193, Green Bay, Wisconsin
  - University of Wisconsin, Site #030, Madison, Wisconsin
- Australia (6):
  - Canberra Hospital, Site #971, Garran, Australian Capital Territory
  - Royal North Shore Hospital, Site #941, Sydney, New South Wales
  - Royal Adelaide Hospital, Site #951, Adelaide, South Australia
  - The Peter MacCallum Cancer Center, Site #950, East Melbourne, Victoria
  - Box Hill Hospital, Site #940, Melbourne, Victoria
  - Royal Perth Hospital, Site #972, Perth, Western Australia
- Medizinische Universitat Wien / AKH, Universitatsklinik fur Inniere Medizin I, Site #561, Vienna, Austria
- Belgium (4):
  - Clinique Universitaire de Saint-Luc, Department of Haematology, Site #508, Brussels
  - UZ Brussel - Department Hematology, Site #544, Brussels
  - UZ Gent - Department Hematology, Site #756, Ghent
  - UZ Gasthuisberg - Department of Hematology, Site #700, Leuven
- Canada (2):
  - University Health Network, Princess Margaret Hospital, Site #083, Toronto, Ontario
  - Jewish General Hospital, Site #129, Montreal, Quebec
- Czechia (4):
  - Fakultni nemocnice Brno, Interni hematologicka a onkologicka klinika, Site #514, Brno
  - FN Hradec Kralove, Site #517, Hradec Králové
  - Fakultni nemocnice Olomouc, Hematoonkologicka klinika, Site #515, Olomouc
  - Ustav hematologie a krevni transfuse, Site #516, Prague
- Helsinki University Central Hospital, Site #542, Helsinki, Finland
- France (14):
  - Institut Bergonie, Site #772, Bordeaux
  - CHRU de Brest, Hopital Morvan, Site #523, Brest
  - CHU Henri Mondor, Site #520, Créteil
  - Centre Hospitalier de Versailles, Site #958, Le Chesnay
  - Hospital Claude Huriez, Site #952, Lille
  - Institut Paoli Calmette, Site #519, Marseille
  - CHU de Brabois, Site #953, Nancy
  - CHU de Nantes, Site #521, Nantes
  - Service Hematologie - Hospital Archet I, Site #509, Nice
  - Hopital Saint-Louis, Site #957, Paris
  - Hospital Saint Antoine, Site #518, Paris
  - Centre Hospitalier Lyon Sud, Site #956, Pierre-Bénite
  - CHU de Poitiers, Site #954, Poitiers
  - CHU Purpan, Site #955, Toulouse
- Germany (9):
  - Universitätsklinikum Aachen, AÖR, Site #513, Aachen
  - Charite - Universitatsmedizin Berlin, Site #701, Berlin
  - Universitatsklinikum Koln-AOR, Site #525, Cologne
  - Universitatsklinikum Carl Gustav Carus an der TU Dresden, Site #526, Dresden
  - Universitatsklinikum Freiburg, Site #527, Freiburg im Breisgau
  - Universitatsklinikum Hamburg-Eppendorf, Site #524, Hamburg
  - Universitatsklinikum Jena, Site #946, Jena
  - Universitat Heidelberg, CML - Studienzentrale III. Medizinische Klinik, Site #947, Mannheim
  - Klinikum rechts der Isar, Site #949, München
- Hong Kong (2):
  - Prince of Wales Hospital, Site #974, Hong Kong
  - Queen Mary Hospital, Site #973, Hong Kong
- Italy (12):
  - Unita Operativa di Ematologia con Trapianto, Site #529, Bari
  - Istituto di Ematologia "L. & A. Seragnoli", Site #959, Bologna
  - A.O. Universitaria Policlinico Vittorio Emanuele di Catania, Site #530, Catania
  - Clinica Ematologica, Site #528, Genova
  - Ospedale Niguarda Ca' Granda di Milano, Site #531, Milan
  - S.C. Ematologia, Site #960, Modena
  - San Gerardo Hospital, Site #961, Monza
  - U.O.C Ematologia con trapianto di midollo osseo, Site #560, Napoli
  - Universita Federico II, Site #510, Napoli
  - SCDU Medicina Interna II - Indirizzo Ematologico, Site #785, Orbassano
  - Dipartimento di Biotecnologie Cellulari ed Ematologia Universita La Sapienza - Policlinico Umberto I, Site #511, Rome
  - U.O. di Ematologia - Ospedale S. Eugenio, Site #962, Rome
- VU Medical Centre - Department Haematology, Site #948, Amsterdam, Netherlands
- New Zealand (4):
  - Auckland City Hospital, Site #921, Grafton, Auckland
  - Christchurch Hospital, Site #922, Christchurch
  - Waikato Hospital, Site #977, Hamilton
  - North Shore Hospital, Site #976, Takapuna
- Poland (5):
  - Klinika Hematologii i Transplantologii, Uniwersyteckie Centrum Medyczne, Site #548, Gdansk
  - Malopolskie Centrum Medyczne, Site #546, Krakow
  - Klinika Hematologii Wojewodzkiego Szpitala Specjalistycznego, Site #550, Lodz
  - Oddzial Hematologii, Site #551, Rzeszów
  - Katedra i Klinika Hematologii, Site #547, Wroclaw
- Instituto Portugues de Oncologia, Site #545, Lisbon, Portugal
- Fundacion de Investigacion de Diego, Site #199, San Juan, Puerto Rico
- Singapore General Hospital, Site #939, Singapore, Singapore
- Slovakia (2):
  - Narodny onkologicky ustav, Site #532, Bratislava
  - Univerzitna nemocnica Martin, Site #533, Martin
- The Catholic University of Korea, Site #938, Seocho-gu, Seoul, South Korea
- Spain (13):
  - Complejo Hospitalario Universitario A Coruna, Hospital "Teresa Herrera," Site #554, A Coruña
  - Hospital Universitari Germans Trias i Pujol, Site #512, Badalona
  - Hospital Clinic, Site #963, Barcelona
  - Institut Catala d' Oncologia de Girona, S. de Hematologia Clinica, Site #734, Girona
  - Hospital Universitari Son Espases, Site #553, Islas Baleares
  - Hospital Universitario La Princesa, Site #555, Madrid
  - Hospital Gregorio Maranon, Site #536, Madrid
  - H.U. Ramon y Cajal, Site #538, Madrid
  - Hospital Universitario 12 de Octubre, Site #537, Madrid
  - Hospital La Paz, Site #966, Madrid
  - Hospital Universitario Central de Asturias, Site #535, Oviedo
  - Hospital Universitario de Salamanca, Site #965, Salamanca
  - Hospital Clinico Universitario de Valencia, Site #964, Valencia
- Sweden (4):
  - Skane University Hospital, Site #944, Lund
  - Karolinska University Hospital Huddinge, Site #534, Stockholm
  - Karolinska University Hospital Solna, Site #763, Stockholm
  - Uppsala University Hospital, Site #945, Uppsala
- Switzerland (2):
  - Kantonsspital Aarau, Site #541, Aarau
  - Kantonsspital St. Gallen, Site #707, Sankt Gallen
- Taiwan (3):
  - Kaohsiung Chang Gung Memorial Hospital, Site #980, Kaohsiung City
  - China Medical University Hospital, Site #978, Taiching
  - National Taiwan University Hospital, Site #979, Taipei
- United Kingdom (10):
  - Western General Hospital, Site #556, Edinburgh
  - Kent and Medway Cancer Research Network, Site #558, Gillingham
  - University of Glasgow, Site #797, Glasgow
  - St. James University Hospital, Site #540, Leeds
  - Royal Liverpool University Hospital, Site #969, Liverpool
  - Hammersmith Hospital, Site #967, London
  - Newcastle University, Site #970, Newcastle
  - Norfolk & Norwich University Hospital Foundation Trust, Site #557, Norwich
  - Nottingham University Hospitals NHS Trust, Site #968, Nottingham
  - Oxford University Hospitals NHS Trust, Site #543, Oxford

REFERENCES:
- [Derived] Hanley MJ, Diderichsen PM, Narasimhan N, Srivastava S, Gupta N, Venkatakrishnan K. Population Pharmacokinetics of Ponatinib in Healthy Adult Volunteers and Patients With Hematologic Malignancies and Model-Informed Dose Selection for Pediatric Development. J Clin Pharmacol. 2022 Apr;62(4):555-567. doi: 10.1002/jcph.1990. Epub 2021 Dec 16. PMID 34699069
- [Derived] Lipton JH, Chuah C, Guerci-Bresler A, Rosti G, Simpson D, Assouline S, Etienne G, Nicolini FE, le Coutre P, Clark RE, Stenke L, Andorsky D, Oehler V, Lustgarten S, Rivera VM, Clackson T, Haluska FG, Baccarani M, Cortes JE, Guilhot F, Hochhaus A, Hughes T, Kantarjian HM, Shah NP, Talpaz M, Deininger MW; EPIC investigators. Ponatinib versus imatinib for newly diagnosed chronic myeloid leukaemia: an international, randomised, open-label, phase 3 trial. Lancet Oncol. 2016 May;17(5):612-21. doi: 10.1016/S1470-2045(16)00080-2. Epub 2016 Apr 12. PMID 27083332

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 307 subjects were enrolled (ponatinib patients: 155; imatinib patients: 152). Patients were randomized in a 1:1 fashion to receive either ponatinib or imatinib.
Period: Overall Study
Arm/Group | Ponatinib | Imatinib
Started | 155 (Started means patient has been randomized.) | 152
Completed | 154 (Completed means patient initiated and discontinued study treatment.) | 152
Not Completed | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Population: ITT Population
Groups:
- Total: Total of all reporting groups
Arm/Group | Ponatinib | Imatinib | Total
Number analyzed (Participants) | 155 | 152 | 307
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 119 | 116 | 235
  >=65 years | 36 | 36 | 72
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.9 (15.66) | 51.2 (15.19) | 51.5 (15.41)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 58 | 60 | 118
  Male | 97 | 92 | 189
Region of Enrollment [Number; unit: participants]
  Portugal | 0 | 2 | 2
  United States | 48 | 34 | 82
  Hong Kong | 4 | 1 | 5
  Taiwan | 3 | 2 | 5
  Finland | 1 | 0 | 1
  Spain | 16 | 9 | 25
  Italy | 15 | 14 | 29
  United Kingdom | 6 | 12 | 18
  France | 14 | 21 | 35
  Czech Republic | 1 | 3 | 4
  Canada | 16 | 13 | 29
  Poland | 0 | 1 | 1
  Belgium | 3 | 2 | 5
  Singapore | 1 | 11 | 12
  Australia | 1 | 6 | 7
  Netherlands | 1 | 1 | 2
  Germany | 11 | 12 | 23
  New Zealand | 4 | 4 | 8
  Sweden | 6 | 2 | 8
  Korea, Republic of | 3 | 2 | 5
  Switzerland | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Major Molecular Response (MMR) Rate at 12 Months
Description: A ratio of reverse transcribed transcript of BCR-ABL to ABL ≤ 0.1% on the international scale, measured by real-time quantitative polymerase chain reaction.
Time Frame: 12 months after first dose
Population: Patients with 12 month assessment (due to early termination of the study, none of the endpoints could be evaluated as planned).
Measure: Number; unit: participants
Arm/Group | Ponatinib | Imatinib
Number analyzed (Participants) | 10 | 13
participants | 8 | 5
Statistical Analysis 1: Comparison: Ponatinib vs Imatinib; Test type: Superiority or Other; p = 0.074, Cochran-Mantel-Haenszel; Stratified Analysis by Sokal score

2. Secondary Outcome: MMR Rate
Description: To compare the efficacy of ponatinib with imatinib, as measured by MMR rate, at 5 years
Time Frame: 5 years after first dose
Reporting Status: Not Posted

3. Secondary Outcome: <10% BCR-ABL^IS Rate
Description: To compare the proportion of patients achieving a ratio of <10% BCR-ABL to ABL transcript levels at 3 months, as measured by the international scale (<10% BCR-ABL^IS), in patients administered ponatinib versus those administered imatinib
Time Frame: 3 months after first dose
Population: Patients with 3 month assessment
Measure: Number; unit: participants
Arm/Group | Ponatinib | Imatinib
Number analyzed (Participants) | 109 | 114
participants | 103 | 77
Statistical Analysis 1: Comparison: Ponatinib vs Imatinib; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel; Stratified Analysis by Sokal score

4. Secondary Outcome: Complete Cytogenetic Response (CCyR) Rate
Description: The percentage of Ph+ metaphases in bone marrow (peripheral blood may not be used), with a review of a minimum of 20 metaphases. Responses are defined as follows: Complete (CCyR): 0% Ph+ metaphases.
Time Frame: 12 months after first dose
Population: Patients with 12 month assessment
Measure: Number; unit: participants
Arm/Group | Ponatinib | Imatinib
Number analyzed (Participants) | 5 | 7
participants | 5 | 6
Statistical Analysis 1: Comparison: Ponatinib vs Imatinib; Test type: Superiority or Other; p = 0.317, Cochran-Mantel-Haenszel; Stratified Analysis by Sokal score

5. Secondary Outcome: Progression-free Survival
Description: To compare, according to treatment with ponatinib versus imatinib, progression-free survival
Time Frame: Up to 8 years after the last patient's first dose
Reporting Status: Not Posted

6. Secondary Outcome: Overall Survival
Description: To compare, according to treatment with ponatinib versus imatinib, overall survival
Time Frame: Up to 8 years after the last patient's first dose
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Patients were followed-up for AEs from the time of informed consent until 30 days after the close of the trial. The median follow-up was 4.97 months (range: 0.03, 17.57) for ponatinib patients, and 5.32 months (range: 0.49, 14.05) for imatinib patients.
Groups:
- Ponatinib 45 mg: ponatinib: 45 mg tablet, taken orally once daily
- Imatinib 400 mg: imatinib (Gleevec/ Glivec): 400 mg tablet, taken orally once daily
Arm/Group | Ponatinib 45 mg | Imatinib 400 mg
Serious Adverse Events (participants affected / at risk) | 49/154 | 13/152
Other Adverse Events (participants affected / at risk) | 145/154 | 144/152
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ponatinib 45 mg (N=154) | Imatinib 400 mg (N=152)
ACUTE MYOCARDIAL INFARCTION (Cardiac disorders) | 2 (2) | 0 (0)
ANGINA PECTORIS (Cardiac disorders) | 2 (2) | 0 (0)
ATRIAL FIBRILLATION (Cardiac disorders) | 3 (3) | 0 (0)
CARDIAC ARREST (Cardiac disorders) | 0 (0) | 1 (1)
CARDIAC FAILURE (Cardiac disorders) | 2 (4) | 0 (0)
CORONARY ARTERY DISEASE (Cardiac disorders) | 1 (1) | 0 (0)
MYOPERICARDITIS (Cardiac disorders) | 1 (1) | 0 (0)
PERICARDIAL EFFUSION (Cardiac disorders) | 1 (1) | 0 (0)
VERTIGO POSITIONAL (Ear and labyrinth disorders) | 1 (1) | 1 (1)
EYE PAIN (Eye disorders) | 1 (1) | 0 (0)
PHOTOPHOBIA (Eye disorders) | 1 (1) | 0 (0)
RETINAL VEIN THROMBOSIS (Eye disorders) | 1 (1) | 0 (0)
ABDOMINAL PAIN (Gastrointestinal disorders) | 2 (3) | 0 (0)
NAUSEA (Gastrointestinal disorders) | 1 (1) | 0 (0)
PANCREATITIS (Gastrointestinal disorders) | 5 (5) | 0 (0)
SMALL INTESTINAL OBSTRUCTION (Gastrointestinal disorders) | 1 (1) | 0 (0)
VOMITING (Gastrointestinal disorders) | 1 (1) | 0 (0)
NON-CARDIAC CHEST PAIN (General disorders) | 1 (1) | 0 (0)
OEDEMA PERIPHERAL (General disorders) | 0 (0) | 1 (2)
PYREXIA (General disorders) | 2 (2) | 1 (1)
SYSTEMIC INFLAMMATORY RESPONSE SYNDROME (General disorders) | 1 (1) | 0 (0)
CHOLECYSTITIS (Hepatobiliary disorders) | 1 (1) | 0 (0)
HEPATITIS (Hepatobiliary disorders) | 0 (0) | 1 (1)
BACTERIAL PYELONEPHRITIS (Infections and infestations) | 1 (1) | 0 (0)
CERVICITIS (Infections and infestations) | 1 (1) | 0 (0)
DISSEMINATED TUBERCULOSIS (Infections and infestations) | 1 (1) | 0 (0)
DIVERTICULITIS (Infections and infestations) | 1 (1) | 0 (0)
HEPATITIS B (Infections and infestations) | 0 (0) | 1 (1)
HERPES ZOSTER (Infections and infestations) | 0 (0) | 1 (1)
LUNG INFECTION (Infections and infestations) | 0 (0) | 1 (1)
PARAINFLUENZAE VIRUS INFECTION (Infections and infestations) | 1 (1) | 0 (0)
PARASPINAL ABSCESS (Infections and infestations) | 0 (0) | 1 (1)
PERICOLIC ABSCESS (Infections and infestations) | 1 (1) | 0 (0)
PNEUMONIA (Infections and infestations) | 2 (3) | 1 (1)
PYELONEPHRITIS (Infections and infestations) | 1 (1) | 0 (0)
RESPIRATORY TRACT INFECTION (Infections and infestations) | 1 (1) | 0 (0)
SEPSIS (Infections and infestations) | 1 (1) | 0 (0)
VESTIBULAR NEURONITIS (Infections and infestations) | 1 (1) | 0 (0)
VIRAL UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 0 (0) | 1 (1)
COMPRESSION FRACTURE (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
PERIORBITAL CONTUSION (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
SPLENIC RUPTURE (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 1 (1) | 0 (0)
AMYLASE INCREASED (Investigations) | 1 (1) | 0 (0)
C-REACTIVE PROTEIN INCREASED (Investigations) | 1 (1) | 0 (0)
PLATELET COUNT DECREASED (Investigations) | 3 (3) | 0 (0)
DECREASED APPETITE (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
FAILURE TO THRIVE (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
HYPONATRAEMIA (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
BONE PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
MUSCULOSKELETAL CHEST PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
NECK PAIN (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
POLYARTHRITIS (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
SACROILIITIS (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
ANGIOMYOLIPOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
BLAST CRISIS IN MYELOGENOUS LEUKAEMIA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
CHLOROMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
CLEAR CELL RENAL CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
CEREBROVASCULAR ACCIDENT (Nervous system disorders) | 1 (1) | 0 (0)
DYSARTHRIA (Nervous system disorders) | 1 (1) | 0 (0)
HEADACHE (Nervous system disorders) | 1 (1) | 0 (0)
HYPOXIC-ISCHAEMIC ENCEPHALOPATHY (Nervous system disorders) | 0 (0) | 1 (1)
LOSS OF CONSCIOUSNESS (Nervous system disorders) | 1 (1) | 0 (0)
POLYNEUROPATHY (Nervous system disorders) | 1 (1) | 0 (0)
PRESYNCOPE (Nervous system disorders) | 0 (0) | 1 (1)
RADICULITIS CERVICAL (Nervous system disorders) | 1 (1) | 0 (0)
TRANSIENT ISCHAEMIC ATTACK (Nervous system disorders) | 1 (1) | 0 (0)
BENIGN PROSTATIC HYPERPLASIA (Reproductive system and breast disorders) | 1 (1) | 0 (0)
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
PLEURAL EFFUSION (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
PULMONARY OEDEMA (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
HYPERTENSION (Vascular disorders) | 1 (1) | 0 (0)
PERIPHERAL ARTERIAL OCCLUSIVE DISEASE (Vascular disorders) | 2 (2) | 0 (0)
PERIPHERAL ARTERY THROMBOSIS (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ponatinib 45 mg (N=154) | Imatinib 400 mg (N=152)
ANAEMIA (Blood and lymphatic system disorders) | 13 (15) | 12 (14)
DRY EYE (Eye disorders) | 10 (10) | 3 (3)
EYELID OEDEMA (Eye disorders) | 1 (1) | 13 (13)
PERIORBITAL OEDEMA (Eye disorders) | 1 (1) | 33 (37)
ABDOMINAL DISCOMFORT (Gastrointestinal disorders) | 10 (11) | 5 (5)
ABDOMINAL PAIN (Gastrointestinal disorders) | 54 (69) | 15 (15)
CONSTIPATION (Gastrointestinal disorders) | 41 (48) | 3 (3)
DIARRHOEA (Gastrointestinal disorders) | 20 (28) | 41 (54)
DRY MOUTH (Gastrointestinal disorders) | 11 (11) | 5 (5)
DYSPEPSIA (Gastrointestinal disorders) | 7 (7) | 9 (10)
NAUSEA (Gastrointestinal disorders) | 34 (44) | 52 (58)
VOMITING (Gastrointestinal disorders) | 17 (18) | 28 (30)
ASTHENIA (General disorders) | 6 (6) | 12 (14)
CHILLS (General disorders) | 10 (12) | 6 (6)
FATIGUE (General disorders) | 32 (37) | 30 (35)
OEDEMA PERIPHERAL (General disorders) | 14 (15) | 22 (24)
PAIN (General disorders) | 9 (10) | 2 (2)
PYREXIA (General disorders) | 26 (31) | 6 (8)
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 5 (5) | 13 (16)
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 20 (29) | 2 (3)
AMYLASE INCREASED (Investigations) | 14 (20) | 1 (1)
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 18 (24) | 6 (7)
BLOOD ALKALINE PHOSPHATASE INCREASED (Investigations) | 14 (20) | 5 (5)
LIPASE INCREASED (Investigations) | 41 (68) | 11 (13)
NEUTROPHIL COUNT DECREASED (Investigations) | 8 (15) | 17 (34)
PLATELET COUNT DECREASED (Investigations) | 36 (65) | 21 (37)
WEIGHT DECREASED (Investigations) | 9 (11) | 2 (2)
WHITE BLOOD CELL COUNT DECREASED (Investigations) | 5 (5) | 9 (11)
DECREASED APPETITE (Metabolism and nutrition disorders) | 18 (20) | 7 (8)
HYPERTRIGLYCERIDAEMIA (Metabolism and nutrition disorders) | 13 (14) | 7 (8)
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 29 (33) | 23 (29)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 11 (13) | 6 (7)
BONE PAIN (Musculoskeletal and connective tissue disorders) | 13 (19) | 12 (16)
MUSCLE SPASMS (Musculoskeletal and connective tissue disorders) | 11 (12) | 52 (62)
MUSCULOSKELETAL PAIN (Musculoskeletal and connective tissue disorders) | 10 (11) | 4 (4)
MYALGIA (Musculoskeletal and connective tissue disorders) | 40 (44) | 27 (31)
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 19 (19) | 12 (15)
DIZZINESS (Nervous system disorders) | 15 (21) | 9 (11)
HEADACHE (Nervous system disorders) | 50 (61) | 20 (27)
LETHARGY (Nervous system disorders) | 3 (3) | 10 (12)
ANXIETY (Psychiatric disorders) | 8 (8) | 5 (5)
DEPRESSION (Psychiatric disorders) | 8 (8) | 5 (5)
INSOMNIA (Psychiatric disorders) | 16 (17) | 4 (4)
COUGH (Respiratory, thoracic and mediastinal disorders) | 8 (9) | 8 (8)
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 13 (18) | 5 (5)
OROPHARYNGEAL PAIN (Respiratory, thoracic and mediastinal disorders) | 10 (10) | 3 (3)
ALOPECIA (Skin and subcutaneous tissue disorders) | 17 (17) | 8 (8)
DRY SKIN (Skin and subcutaneous tissue disorders) | 27 (29) | 5 (5)
ERYTHEMA (Skin and subcutaneous tissue disorders) | 11 (12) | 2 (3)
NIGHT SWEATS (Skin and subcutaneous tissue disorders) | 7 (7) | 9 (10)
PRURITUS (Skin and subcutaneous tissue disorders) | 18 (20) | 11 (15)
RASH (Skin and subcutaneous tissue disorders) | 58 (100) | 25 (41)
RASH PRURITIC (Skin and subcutaneous tissue disorders) | 6 (8) | 11 (14)
HYPERTENSION (Vascular disorders) | 27 (37) | 3 (4)

LIMITATIONS AND CAVEATS:
Trial was discontinued early.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No